CLINICAL TRIAL: NCT05745012
Title: Anti-Reflux Mucosectomy (ARMS) in the Treatment of Refractory Gastro-esophageal Reflux (GERD): a Prospective Randomized Comparative Study
Brief Title: Anti-Reflux Mucosectomy in the Treatment of Refractory Gastro-esophageal Reflux
Acronym: MARRGO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-A00599-34
Record Dates: First submitted 2022-09-05; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Gastroesophageal Reflux Disease With Ulceration
MeSH Terms: interventions — Endoscopic Mucosal Resection; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: operating gastroenterologist will be unblind while evaluating gastroenterologist will be blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A: control group (Sham Comparator)
  Interventions: Procedure: sham
- group B: ARMS procedure (Experimental)
  Interventions: Procedure: endoscopic mucosal resection

INTERVENTIONS:
Procedure: endoscopic mucosal resection — The procedure consists of performing endoscopic mucosal resection of the 3/4 of the circumference of the esogastric junction using the Duette system (Cook Endoscopy, USA). The procedure will be performed under general anesthesia in an intubated patient, and realized in ambulatory setting.
  Arms: group B: ARMS procedure
Procedure: sham — The procedure consists of performing endoscopic exploration, no mucosal resection
  Arms: group A: control group

SUMMARY:
Gastroesophageal reflux disease (GERD) is one of the most common digestive diseases in Western countries, affecting 8% of the population in its typical and frequent form. For typical GERD without alarming symptoms, treatment combines PPI therapy and lifestyle modifications. Patients with an incomplete response to optimized PPI therapy have so-called refractory GERD. Anti-reflux mucosectomy (ARMS) is a recent technique that achieves endoscopic fundoplication by scar-induced tissue retraction using a mucosal ligation system combined with resection, known as the banded ligation system (ARM-b) [6]. Several studies have shown efficacy of approximately 65-70% on symptom resolution and quality of life improvement, including our pilot study of 21 patients, and without serious adverse events.

The purpose of this study is therefore to prospectively evaluate in a randomized blinded comparison to a sham procedure and conventional medical follow-up, the efficacy of anti-reflux mucosectomy (ARMS) in the treatment of refractory GERD.

The hypothesis is that we can achieve a clinical efficacy rate of 65% in the treatment group versus 35% in the control group.

The primary objective is to demonstrate the superiority in terms of clinical efficacy (self-reported symptom-related GERD rate, GERD-SLR) of RAS compared to the sham procedure combined with optimized medical treatment at 1 year. The primary endpoint will be clinical efficacy, defined as a greater than 50% decrease in the number of GERD-associated symptoms, assessed using the GERD-HRQL score.

Secondary objectives will be:

Assessing clinical efficacy at 6 months. Assess the impact on PPI use Assess changes in procedure-induced abnormal esophageal acid exposure by Ph-metry Assess the impact of this technique on patient quality of life; To document the adverse effects of the technique (AGREE, Clavien Dindo and ASGE score) The duration of follow-up will be 1 year, and based on our hypothesis the number of patients to be included will be 130.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient that have read the information form and signed consent
* Patient covered with health insurance
* GERD with typical symptom of pyrosis, or atypical symptoms with clinical symptomatic correlation confirmed by pre-operative Ph-Impedencemetry performed in the last 6 months
* GERD evolving for at least 1 year, and refractory to medical treatment, which is defined by the persistence of daily GERD related symptoms despite PPI at 20mg twice daily associated with local topics and hygiene-dietary measures
* High-resolution manometry (HRM) to eliminate severe motor disorder and research lower esophageal sphincter hypotony performed in the last 6 months
* Eso-gastro-duodenoscopy (EGD) to confirm the absence of severe esophagitis, hiatal hernia, and complicated Barret's esophagus performed in the last 3 months

Exclusion Criteria:

* Grade C peptic esophagitis (Los Angeles classification), persisting despite medical treatment at pre-inclusion gastroscopy (< 6 months)
* Hiatal hernia > 2cm at preoperative gastroscopy
* Barret's Esophagus > C0-M2 with relief abnormalities or confirmed high-grade dysplasia (2 endoscopies within 6 months)
* History of esophageal or gastric surgery
* Severe esophageal motility disorder at HRM such as achalasia or spastic disorder (Chicago classification); minor motility disorders may be included
* No french language comprehension
* Patient under tutelle or curatelle
* Patient already enrolled in interventional research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
demonstrate superiority of ARMS | one year
  the clinical efficacy defined as the decreasing of self-reported related-symptom GERD assessed using the GERD-HRQL score of more than 50% at one year

SECONDARY OUTCOMES:
Assessing the clinical efficacy at 6 months | 6 months
  The clinical efficacy, as defined above, at 6 months
Evaluating the impact on PPIs use after ARMS and sham procedures, respectively; | one year
  The rate (and the date) of complete disruption of PPIs at 1 year if so, or, in case of decreasing the mean daily or weekly dose compared to before the intervention
Assessing the changes in abnormal exposure to esophageal acid induced by the procedure | 3 months
  The % time with Ph under 4 on post-operative (3 months) Ph-impedencemetry, compared to pre-operative
Assessing the changes in abnormal exposure to esophageal acid induced by the procedure | 3 months
  the De Meester score. The interpretation of the score is as follows:
  * DMS <14.72 No GERD
  * DMS 14.72 - 50 Mild GERD
  * DMS 51 - 100 Moderate GERD
  * DMS >100 Severe GERD
Evaluating the impact of this technique on patients' quality of life; | 2 months
  The quality of life based on Gastrointestinal Quality of Life index (GIQLI) at 2 months These scores are validated to assess the quality of life specific to digestive diseases. They are free of used and traduced in French. there is no report on a scale
Evaluating the impact of this technique on patients' quality of life; | 4 months
  The quality of life based on Gastrointestinal Quality of Life index (GIQLI) at 4 months These scores are validated to assess the quality of life specific to digestive diseases. They are free of used and traduced in French. there is no report on a scale
Evaluating the impact of this technique on patients' quality of life; | 6 months
  The quality of life based on Gastrointestinal Quality of Life index (GIQLI) at 6 months. These scores are validated to assess the quality of life specific to digestive diseases. They are free of used and traduced in French. there is no report on a scale
Evaluating the impact of this technique on patients' quality of life; | one year
  The quality of life based on Gastrointestinal Quality of Life index (GIQLI) at 1 year. These scores are validated to assess the quality of life specific to digestive diseases. They are free of used and traduced in French. there is no report on a scale
Evaluating the impact of this technique on patients' quality of life; | 2 months
  The quality of life based on SF12 scores at 2 months. These scores are validated to assess the quality of life specific to digestive diseases. They are free of used and traduced in French. there is no report on a scale
Evaluating the impact of this technique on patients' quality of life; | 4 months
  The quality of life based on SF12 scores at 4 months. These scores are validated to assess the quality of life specific to digestive diseases. They are free of used and traduced in French. there is no report on a scale
Evaluating the impact of this technique on patients' quality of life; | 6 months
  The quality of life based on SF12 scores at 6 months. These scores are validated to assess the quality of life specific to digestive diseases. They are free of used and traduced in French. there is no report on a scale
Evaluating the impact of this technique on patients' quality of life; | one year
  The quality of life based on SF12 scores at 1 year. These scores are validated to assess the quality of life specific to digestive diseases. They are free of used and traduced in French. there is no report on a scale
Documenting the adverse events of the technique; | one year
  The adverse events rate of ARMS procedure, evaluated per-operatively and until 30 post-operative days, their severity assessed using the AGREE classification, and their management

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HM, Marseille, France

IPD SHARING:
Plan to Share IPD: No